CLINICAL TRIAL: NCT01873183
Title: Perioperative Fluid Management With Transthoracic Echocardiography and Pulse-contour Device in Morbidly Obese Patients
Brief Title: Perioperative Fluid Management in Morbidly Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Tomi Myrberg, Senior lecturer, MD PhD, Umeå University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-439-32M
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Hypotension; Anomaly; Venous Return; Dehydration
Keywords: echocardiography; morbid obesity; bariatric surgery; venous return; mean arterial blood pressure
MeSH Terms: conditions — Hypotension; Congenital Abnormalities; Dehydration; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The IGDT group (Experimental): 30 morbidly obese subjects scheduled for bariatric surgery by laparoscopic Roux-en-Y gastric bypass (RYGB) will be consecutively enrolled for the study.
  The individualized goal-directed therapy (IGDT) with focus on level of venous return will be implemented in two steps in the intervention group. First, preoperative optimizing of venous return will be performed 45 minutes before surgery in a preoperative room with TTE. Second, after induction of anaesthesia perioperative fluid therapy will be implemented by utilizing the FloTrac-device.
  Interventions: Other: Goal directed fluid therapy
- The control group (No Intervention): 20 morbidly obese subjects scheduled for bariatric surgery by laparoscopic Roux-en-Y gastric bypass (RYGB) will consecutively be enrolled for the study. Conventional monitoring will be conducted perioperatively.

INTERVENTIONS:
Other: Goal directed fluid therapy
  Arms: The IGDT group

SUMMARY:
In bariatric surgery functional and feasible non- or mini-invasive modalities for monitoring, and ideal/lean body weight estimates are addressed to meet up individual variability in hydration needs, and to avoid hyperhydration.

The aim of the study is to evaluate need of perioperative hydration by comparing conventional monitoring (the control group) to a more advanced approach (individualized goal-directed therapy, IGDT) (the intervention group). In addition to conventional cardiovascular monitoring (ECG, non-invasive blood pressure, Sp02) preoperative transthoracic echocardiography (TTE) and a intraoperative perioperative mini-invasive pulse-contour device (FloTrac™) will be used for the purpose.

DETAILED DESCRIPTION:
The individualized goal-directed therapy (IGDT), with focus on level of venous return, will be implemented in two steps in the intervention group. First, preoperative optimizing of venous return will be performed 45 minutes before surgery in a preoperative room with TTE. Second, after induction of anaesthesia perioperative fluid therapy will be guided by utilizing the FloTrac-device.

Preoperative rehydration with 6 ml colloid fluids (Volulyte™, Fresenius Kabi Ab, Sweden) /kg estimated ideal body weight (IBW) will be administrated if low level of venous return is detected by TTE. After a colloid bolus the second TTE is performed to check the level of venous return. If remaining hypovolemia is found additional colloids 3ml/ kg IBW will be given.

In OR, before pneumoperitoneum, prophylactic i.v. antibiotics will be administrated in total 550ml crystalloids (NaCl 0.9%, Fresenius Kabi Ab, Sweden) to all patients. Infusion of buffered glucose solution (25mg/ml, Fresenius Kabi Ab, Sweden) at rate 1.5ml/kg IBW/h will be initiated to all patients. Stroke volume variation ≥ 12 % is used as a threshold for administration of additional colloids 3ml/kg/ IBW during surgery.

Postoperatively infusion of buffered glucose solution (50mg/ml) is administrated at fixed rate 100ml/h to all patients. In addition, during the stay at the postoperative ward unit 850 ml crystalloids (antibiotics, paracetamol and nonsteroidal antiinflammatory drugs) are infused.

Perioperative ephedrine and/or phenylephrine is used as i.v. injection when necessary to ensure adequate perfusion pressure (MAP ≥ 65 mmHg), cardiac index (≥ 2.0) and heart rate (≥ 50/min) in addition to i.v. fluids in both groups. In principle hemodynamic parameters will be gathered always after five minutes minimum from possible administration of i.v. ephedrine or phenylephrine. Moreover, if pre-existing systolic left ventricular failure is detected in preoperative TTE, infusion of dobutamine 3 - 4ug/kg IBW will be started 10 minutes before induction of anaesthesia.

In the control group perioperative cardiovascular monitoring will be conducted by ECG, non-invasive blood pressure and Sp02 measurements.

ELIGIBILITY:
Inclusion Criteria:

* accepted for bariatric surgery; BMI ≥ 40 kg/m2. Written informed consent. Successful preparation by 3 weeks rapid-weight-loss diet before surgery (≥ 5% loss of weight)

Exclusion Criteria:

* Subjects with untreated systemic or pulmonary hypertension, atrial fibrillation, pacemaker, unstable angina pectoris and significant failure of heart valves.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Need of perioperative i.v. fluids | 12 hours
  The primary aim of the study is to evaluate need of perioperative hydration during laparoscopic bariatric surgery. Type and amount of all perioperative fluids infused will be registered. Timing for administration of fluids will be analysed in three steps (preoperative, operating room (OR) and postoperative).

SECONDARY OUTCOMES:
mean arterial blood pressure | 1 hour
  Mean arterial blood pressure (MAP) will be measured before induction of anaesthesia, 5 min after endotracheal intubation, 5 min after deep reverse Trendelenburg position and pneumoperitoneum in the intervention and the control groups. In addition, MAP will be registered continuously during surgery.

OTHER OUTCOMES:
Nt-proBNP, creatinine | 12 hours
  A baseline for Nt-proBNP and creatinine will be taken before i.v fluids preoperatively on the day of surgery. Control samples will be gathered 12 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Tomi P Poso, MD, Principal Investigator — Umea University
Locations (1):
- Department of anaesthesiology and intensive care, Sunderby county hospital, Luleå, Sweden

REFERENCES:
- [Derived] Poso T, Winso O, Aroch R, Kesek D. Perioperative fluid guidance with transthoracic echocardiography and pulse-contour device in morbidly obese patients. Obes Surg. 2014 Dec;24(12):2117-25. doi: 10.1007/s11695-014-1329-4. PMID 24902655